CLINICAL TRIAL: NCT04182958
Title: A Phase I, Open-Label Trial to Assess the Mass Balance and Pharmacokinetics of a Single Intravenous Administration of (14C)-OPC-61815 to Healthy Male Japanese Subjects
Brief Title: A Phase I, Open-Label Trial to Assess the Absorption, Metabolism, and Excretion of (14C)-OPC-61815 in Healthy Male Japanese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 263-102-00006; 2019-001968-29 (EudraCT Number)
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Results first posted 2021-10-06 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Healthy Adult Male

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- (14C)-OPC-61815 (Experimental)
  Interventions: Drug: (14C)-OPC-61815

INTERVENTIONS:
Drug: (14C)-OPC-61815 — On the morning of Day 1, all subjects will receive a single IV infusion of (14C) OPC-61815

SUMMARY:
* To determine the mass balance of totalradioactivity following a single IV infusionof (14C)-OPC-61815.
* To determine routes and rates of elimination of total radioactivity following a single IV infusion of (14C)-OPC-61815
* To assess the PK of total radioactivity in plasma and whole blood following a single IV infusion of (14C)-OPC-61815
* To assess the PK of OPC-61815 free form and OPC-41061 in plasma following a single IV infusion of (14C)-OPC-61815

ELIGIBILITY:
Inclusion Criteria:

* Male subjects between 35 and 55 years of age, inclusive; hold a valid Japanese passport and be first generation Japanese, defined as the subject, the subject's biological parent, and all of the subject's biological grandparents being of exclusive Japanese descent, have been born in Japan, and not lived outside of Japan for more than 5 years; with a body mass index between 18.5 and 28.0 kg/m2, inclusive, and a total body weight between 50 and 100 kg, inclusive; in good health, determined by no clinically significant findings from medical history, physical examination, 12-lead electrocardiogram (ECG), vital sign measurements, and clinical laboratory evaluations at Screening and Check in as assessed by the investigator (or designee); and have a history of a minimum of 1 bowel movement per day.

Exclusion Criteria:

* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion; poor peripheral venous access; participation in a clinical trial involving administration of an investigational drug in the past 90 days prior to dosing; subjects with exposure to significant diagnostic or therapeutic radiation or current employment in a job requiring radiation exposure monitoring within 12 months prior to Check-in; subjects who have participated in any clinical trial involving a radiolabeled investigational drug within 12 months prior to Check-in.

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takehisa Matsumaru, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Covance Clinical Research Unit Ltd, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Small studies with less than 25 participants are excluded from data sharing.

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall: (14C)-OPC-61815: Subjects were to receive a single IV infusion of 16 mg (14C)-OPC-61815, containing approximately 75.1 μCi (2.78 MBq), over a period of 60 minutes (55 to 65 minutes, inclusive) on Day 1 of the trial.
Period: Overall Study
Arm/Group | Overall: (14C)-OPC-61815
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall: (14C)-OPC-61815
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Japanese | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 8

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUC∞) - Plasma OPC-61815 Free Form
Time Frame: 48 hours after dose
Population: The PK population included all subjects that received (14C)-OPC-61815 (full dose within the time frame of 55 to 65 minutes, inclusive) and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Overall: (14C)-OPC-61815
Number analyzed (Participants) | 8
h*ng/mL | 2060 (305)

2. Primary Outcome: Maximum Peak Concentration (Cmax) - Plasma OPC-61815 Free Form
Time Frame: 48 hours after dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Overall: (14C)-OPC-61815
Number analyzed (Participants) | 8
ng/mL | 1500 (156)

3. Primary Outcome: Terminal-phase Elimination Half-life (t1/2,z) - Plasma OPC-61815 Free Form
Time Frame: 48 hours after dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Overall: (14C)-OPC-61815
Number analyzed (Participants) | 8
hours | 3.61 (1.34)

4. Primary Outcome: AUC∞ - Plasma OPC-41061
Time Frame: 48 hours after dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Overall: (14C)-OPC-61815
Number analyzed (Participants) | 8
h*ng/mL | 1150 (230)

5. Primary Outcome: Cmax - Plasma OPC-41061
Time Frame: 48 hours after dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Overall: (14C)-OPC-61815
Number analyzed (Participants) | 8
ng/mL | 204 (27.9)

6. Primary Outcome: t1/2,z - Plasma OPC-41061
Time Frame: 48 hours after dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Overall: (14C)-OPC-61815
Number analyzed (Participants) | 8
hours | 5.27 (0.826)

7. Primary Outcome: AUC∞ - Plasma Total Radioactivity
Time Frame: 168 hours after dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ngEq/mL
Arm/Group | Overall: (14C)-OPC-61815
Number analyzed (Participants) | 8
h*ngEq/mL | 30300 (4850)

8. Primary Outcome: Cmax - Plasma Total Radioactivity
Time Frame: 168 hours after dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ngEq/mL
Arm/Group | Overall: (14C)-OPC-61815
Number analyzed (Participants) | 8
ngEq/mL | 2180 (188)

9. Primary Outcome: t1/2,z - Plasma Total Radioactivity
Time Frame: 168 hours after dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Overall: (14C)-OPC-61815
Number analyzed (Participants) | 8
hours | 128 (33.1)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from the start of investigational medicinal product (IMP) administration up to 12 days
Description: The safety population included all subjects that received (14C)-OPC-61815.
Arm/Group | Overall: (14C)-OPC-61815
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall: (14C)-OPC-61815 (N=8)
Rash (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/58/NCT04182958/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT04182958/SAP_001.pdf